CLINICAL TRIAL: NCT06393699
Title: Restoration of Non-carious Cervical Lesions: The Effect of Different Resin Composites Bonded With A Universal Adhesive Utilizing Two Adhesion Approaches: A Randomized Clinical Study
Brief Title: Restoration of Non-carious Cervical Lesions With Different Resin Composites and Universal Adhesive
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Aisha Ahmed Elbaz, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 969
Record Dates: First submitted 2023-08-29; First posted 2024-05-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Retention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- incremental (Experimental): application of increments of packable composite in non carious cervical lesions
  Interventions: Procedure: composite restoration
- bulk fill heated (Experimental): application of heated composite as bulk in the lesions without incrementation after heating with caps warmer
  Interventions: Procedure: composite restoration
- incremental heated (Experimental): application of composite in increments after being heated by caps warmer
  Interventions: Procedure: composite restoration
- flowable (Experimental): application of flowable composite in non carious cervical lesions
  Interventions: Procedure: composite restoration

INTERVENTIONS:
Procedure: composite restoration — different types of resin composite restorations will be used to restore NCCL

SUMMARY:
patients with non carious cervical lesions suffer from dentin sensitivity and presence of cavitations and gingival recession. Restoring these lesions with different composites and evaluation of restorations every 6 months will be done to know the effect of different composite types and consistencies in retention of restorations of such lesions.

DETAILED DESCRIPTION:
A split-mouth randomized clinical trial (RCT), based on the adhesion strategy, will be held on 52 patients attending to the outpatient clinics of the department of operative dentistry, Faculty of Dentistry, Ain Shams University with 2 non-carious cervical lesions in each side. Patients included in this study are those who seek restorative treatment of non-carious cervical lesions (NCCLs) in premolars and canines, which are due to chemical and/or mechanical predisposing factors. An informed consent will be signed by all participants who will be allocated in this study before being involved in the study. Male and female patients will be selected according to the inclusion and exclusion criteria. The patients will be randomly assigned into 4 main groups (n=13 patients/group) according to the type of restorative material will be inserted. In each group, two adhesive approaches will be employed, either etch-and-rinse (E&R) or self-etching (SE)approach. For each patient's mouth, one side will receive restorations with the etch-and-rinse approach (n=26 restorations/E&R approach), while the other side will receive restorations using the self-etching approach (n=26 restorations/SE approach). This will result in a total of 208 restorations will be inserted in this study. A treatment follow-up will be performed every six months for two years to investigate the clinical performance of the different resin composite restorations/the two different adhesive approaches.

Restorations will be evaluated at baseline and every 6 months by two blinded examiners, who will not be involved in the study. During evaluation, the examiners will not be informed about the type of restoration used or the adhesive approach and will have a code for each patient and the restored tooth. Restorations will be evaluated according to the modified United State Public Health Service criteria (USPHS).(6,9,13,30) Primary outcome will be the retention of the restoration, but the following secondary outcomes as marginal discoloration and adaptation, anatomic form, secondary caries, texture, and postoperative sensitivity will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

- Patients' age will range from 18 to 65 years.

* Presence of at least 2 NCCLs in one side.
* Patients with no medical condition could interfere with the routine dental care.
* Patients who will be able to attend for each recall visit.
* Patients with healthy periodontal tissues.
* Cavities presenting no more than 50% of margins in enamel.

Exclusion Criteria:

* Medically compromised patients.

  * Pregnant or breast-feeding patients.
  * Patients undergoing orthodontic treatment or bleaching treatment in the time of the study.
  * Patients with periodontal disease in the target area.
  * Patients presented with less than 20 teeth in the oral cavity.
  * Patients without antagonists.
  * Lesions superimposed with caries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-05-14 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Retention | 18-24 months
  ability of resin composite restorations to be retained in the non carious cervical lesions

SECONDARY OUTCOMES:
marginal staining | 18-24 months
  will be assessed visually by blinded evaluator

OTHER OUTCOMES:
Marginal adaptation | 18-24 months
  will be assessed by explorer done by blinded evaluator
postoperative sensitivity | 18-24 months
  will be assessed using triple way syringe with air done by blinded evaluator

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: expecting to have all data by october 2026